CLINICAL TRIAL: NCT03356314
Title: Prenatal Ultrasound Screening of Intestinal Malrotation With a Higher Risk of Volvulus: Value of The Relative Position of The Superior Mesenteric Artery and Vein. Future of the Children With an Antenatal Malrotation Suspicion
Brief Title: Prenatal Ultrasound Screening of Intestinal Malrotation With a Higher Risk of Volvulus
Acronym: VOLMES
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0258
Record Dates: First submitted 2017-10-12; First posted 2017-11-29 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2017-10

CONDITIONS: Intestinal Malrotation
Keywords: superior mesenteric artery; superior mesenteric vein; intestinal malrotation; volvulus; pregnant women; mesenteric vessels position; postnatal diagnosis; prophylactic surgery
MeSH Terms: conditions — Volvulus Of Midgut; Intestinal Volvulus | interventions — Barium Enema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI between 30-35 GA — MRI between 30-35 GA
Other: Pediatric surgeon meeting — Pediatric surgeon meeting
Other: Postnatal abdominal ultrasound, barium enema and upper gastrointestinal — Postnatal abdominal ultrasound, barium enema and upper gastrointestinal
Other: +/- prophylactic surgery — +/- prophylactic surgery

SUMMARY:
The aim of this study was to assess the value of an unusual relative position of the superior mesenteric artery (SMA) and vein (SMV) to screen intestinal malrotation with a higher risk of volvulus.

First, feasibility study was done to prove the reproducibility of ultrasound in diagnosis of anormal mesenteric vessels position.

A systematic screening of the mesenteric vessels position was performed at each pregnancy required ultrasound.

When the fœtus had an unusual position of the mesenteric vessels, an MRI was suggested between 30 and 35 GA and the couple met the pediatric surgery team.

Few days after birth, an abdominal ultrasound was achieved as well as a barium enema and upper gastrointestinal. If there were a hight probability of malrotation with a higher risk of volvulus, a prophylactic surgery was proposed. The children were flollowed up during 1 year.

ELIGIBILITY:
Inclusion criteria:

* pregnant women
* second or third trimester ultrasound.

Exclusion criteria:

* fœtal ultrasound anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pregnant women
Sampling Method: Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Reproducibility of ultrasound in the diagnosis of the abnormal position of the mesenteric vessels | 1 day (Pre and post natal ultrasound)
  Feasibility study to prove the reproducibility of ultrasound in diagnosis of anormal mesenteric vessels position.
Antenatal screening of intestinal malrotation | 1 day (Pre and post natal ultrasound)
  Antenatal screening of intestinal malrotation with higher risk of volvulus.
Future of the children with an ante natal diagnosis of intestinal malrotation | 1 year after birth
  Future of the children with an ante natal diagnosis of intestinal malrotation

SECONDARY OUTCOMES:
Produce ante and postnatal strategy facing a situation of mesenteric vessels malposition. | 1 day (During Pregnancy)
  Produce ante and postnatal strategy facing a situation of mesenteric vessels malposition.
Produce ante and postnatal strategy facing a situation of mesenteric vessels malposition. | 1 day (after delivery)
  Produce ante and postnatal strategy facing a situation of mesenteric vessels malposition.

CONTACTS AND LOCATIONS:
Overall Officials: florent FUCHS, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC